CLINICAL TRIAL: NCT06987357
Title: Comparison of the Effects of Sugammadex and Neostigmine on Early Extubation, Intensive Care Unit Admission and Length of Stay, and Hospital Costs in Adult Cranial Surgery
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Naime Yalçın, Specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.04.116
Record Dates: First submitted 2025-05-09; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Craniectomy; Sugammadex; Extubation; Recovery After Neuromuscular Block; Hospital Costs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Neostigmine
- Group Sugammadex

SUMMARY:
The aim of this study was to retrospectively investigate the effects of sugammadex or neostigmine, which are routinely used after the completion of surgery to antagonize (reverse) neuromuscular blockade in adult patients undergoing cranial surgery under general anesthesia, on early extubation in the operating room, intensive care unit admission and length of stay, length of hospital stay, and hospital costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the American Society of Anesthesiology (ASA) I-II-III group,
* over the age of 18,
* who underwent elective surgery,
* underwent general anesthesia with sevoflurane anesthesia from volatile anesthetics,
* used rocuronium as a neuromuscular blocking agent

Exclusion Criteria:

* Patients aged 18 and under,
* ASA IV and above,
* who underwent surgery under emergency conditions,
* who have incomplete follow-up form records and electronic media data,
* who were taken to the intensive care unit without neuromuscular blockade antagonism due to long surgery,
* who were treated with a neuromuscular blocking agent other than rocuronium,
* who were treated with a volatile anesthetic other than sevoflurane or with total intravenous anesthesia.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients who underwent cranial surgery under sevoflurane anesthesia and whose neuromuscular blockade was provided with rocuronium, the patients whose neuromuscular blockade was antagonized with neostigmine or sugammadex and who were admitted to the intensive care unit postoperatively were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The amount of cost in the hospital process | through study completion, an average of 3 month
Length of stay in the intensive care unit | through study completion, an average of 3 month
Early extubation rate after two different neuromuscular blocking antagonist drugs | through study completion, an average of 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)